CLINICAL TRIAL: NCT03901183
Title: Plant-based Nutrition for Patients With Cardiovascular Risk Factors - a Randomized Controlled Trial
Brief Title: Plant-based Nutrition for Patients With Cardiovascular Risk Factors
Acronym: CardioVeg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Charite University, Department for Dental Medicine (Unknown)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CardioVeg
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Metabolic Syndrome; Cardiovascular Risk Factor; Overweight and Obesity; Hypertension,Essential
Keywords: Metabolic Syndrom; Plant-based Diet; Nutrition
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Obesity; Essential Hypertension | interventions — Diet, Plant-Based

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Participants receive a 8 week nutritional counseling with weekly group meetings to establish a plant-based diet.
  Interventions: Other: Plant-based Diet
- Control (No Intervention): Waiting list. Participants receive no intervention during study period, equal intervention is offered after the end of study.

INTERVENTIONS:
Other: Plant-based Diet — Patients are guided to change their nutrition to a plant-based diet.
  Arms: Interventional

SUMMARY:
Plant-based nutrition may have positive effects on chronic diseases such as cardiovascular or metabolic disorders. This study investigates the effects of a 8 week plant-based diet for patients with metabolic syndrom and cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure > 140 mmHg systolic and/or > 90 mmHg diastolic, in case of medication also increased values > 140 mmHg systolic and/or > 90 mmHg diastolic needed
* Adipositas with a waist circumference of > 94 cm in men and > 80 cm in women
* A non-vegetarian diet in the past 6 months (at least 4x meat and/or meat products per week, at least 5x dairy products per week)
* No fasting, no specific diet or change of diet in the last 2 months
* Weight stable over the last two months (+- 3 kg)
* Medication unchanged for at least one month
* No fasting, no change of diet in the last 2 months

Exclusion Criteria:

* Poor general condition
* Coronary heart disease
* Diabetes mellitus Type I
* Cerebrovascular diseases
* Severe mental illness
* Severe acute or chronic comorbidity
* Pregnancy and lactation or planned pregnancy in the next 6 months
* Eating disorder
* Max. 2 beers 0,5l or 2 wines 0,2l per day
* No alcohol abstinence 48 hours before blood samples possible
* Max. 5 cigarettes/day
* Medicine that affect weight
* Antibiotics within the last 6 months
* Major surgery <6 months prior to randomization
* BMI > 40 kg/m2
* Existing vegetarian or plant-based diet
* Bariatric surgery (obesity surgery)
* Simultaneous participation in another clinical trial
* Participation in a clinical trial within the last 3 months prior to inclusion in the study
* Lack of consent to participate in the study

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Change of baseline Composite Score for Metabolic Syndrom (Standardizing Physiological Composite Risk Endpoints (SCORE)) at 2 months | Date of inclusion (baseline), after 8 weeks
  Composite score including waist wircumference, blood pressure, fasting blood glucose, tryglycerids, HDL-cholesterin Range 0-100, lower score meaning a better outcome

SECONDARY OUTCOMES:
Bio-electrical Impedance Analysis (BIA) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Estimation of the body composition via bio-electrical impedance analysis (body fat and visceral fat in %)
Bio-electrical Impedance analysis (BIA) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Estimation of the body composition via bio-electrical impedance analysis (muscle mass in kg)
Change from baseline systolic blood pressure at 2 months | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Average of 24h measurement
Change from baseline diastolic blood pressure at 2 months | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Average of 24h measurement
Fasting glucose (mmol/l) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
Blood lipids | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Triglycerides (mmol/L), total cholesterol (mmol/L), LDL (mmol/L), HDL (mmol/L)
Insulin (µU/ml) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
Glycated hemoglobin (HbA1c) (%) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
Fructosamin (µmol/l) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
Homeostatic model assessment (HOMA-IR) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Index calculated from Insulin (µU/ml) x fasting glucose (mmol/l) / 22,5
Ferritin (µg/l) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
Liver enzymes | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Hepatic transaminases (GPT, GOT in U/L) and Gamma glutamyl transpeptidase (y-GT in U/L)
Folic acid (ng/ml) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
Uric Acid (mg/dl) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
Complete Blood Count | Date of inclusion (baseline), after 8 weeks, after 16 weeks
Holotranscobalamin (pmol/L) | Date of inclusion (baseline), after 16 weeks
Trimethylamine N-oxide (mg/dl) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
Quality of Life questionnaire (WHO-5) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Change from Baseline in the WHO-5, range from 0 to 100 % while higher values meaning a higher grade of well-being
Stress questionnaire (Cohen Perceived Stress Scale, CPSS) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Change from Baseline in the CPSS, range from 0 to 4 in each item. Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the positively stated items and then summing across all scale items while higher values meaning a higher grade of perceived stress.
General Self-efficacy Short Scale (ASKU) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Assessing full scale, range 3-15, higher score meaning a better outcome
Hospital Anxiety and Depression Scale (HADS) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Assessing full scale, range 0-42, lower score meaning a better outcome
Medical Outcomes Study Short Form (MOS SF-12) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Assessing full scale, range 0-100, higher score meaning a better outcome
Zerssen symptom list (B-LR and B-LR') | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Assessing full scale, range 20-80, higher score meaning a better outcome
Intuitive Eating Scale 2 (IES-2) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Assessing full scale, range 23-115, higher score meaning a better outcome
Flourishing Scale (FS-D) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Assessing full scale, range 8-56, higher score meaning a better outcome
International Physical Activity Questionnaire (IPAQ ) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  MET minutes represent the amount of energy expended carrying out physical activity. To get a continuous variable score from the IPAQ (MET minutes a week) we will consider walking to be 3.3 METS, moderate physical activity to be 4 METS and vigorous physical activity to be 8 METS.
Body weight (kg) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
Body Mass Index (kg/m2) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
Waist circumference (cm) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
Wrist Circumference (cm) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
Ambulatory Blood Pressure Monitoring (ABPM) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Measuring systolic and diastolic blood pressure in 20-minute-intervals for 24h with "Spacelabs" devices
Dietary Behaviour | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Nutritional history via dietary weight record (each for 3 days)
Daily nutrition protocol | Daily throughout the entire survey period
  Via the App 'Calorie Counter - Fddb Extender'
Medication intake | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Name of medication and dosage
Cardio Vascular Risc Profile | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Cardio Vascular Risc in % with following scores: SCORE-Deutschland/PROCAM/arriba/WHO-ISH Charts/BEWAT-Score
Gut microbiome | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  16S rRNA Sequencing / Shotgun Sequencing
Blood Oxygenization | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by Biovotion Everion (upper arm)
Skin Temperature | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by Biovotion Everion and Empatica E4 devices (upper arm/wrist)
Heart Rate (HR) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by Faros 180 (chest), Biovotion Everion and Empatica E4 (upper arm/wrist) devices
Heart Rate Variability (HRV) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by Faros 180 (chest), Biovotion Everion and Empatica E4 (upper arm/wrist) devices
Interbeat Interval (IBI) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by Biovotion Everion and Empatica E4 devices (upper arm/wrist)
Respiration Rate | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by Biovotion Everion device
Blood Volume Pulse | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by Empatica E4 device (wrist)
Electrodermal Activity (Galvanic Skin Response) | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by Biovotion Everion device and Empatica E4 (upper arm/wrist) devices
Number of Steps per 24 hours | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  24h measuring by Biovotion Everion device (upper arm)
Sociodemographic Measurements | Date of inclusion (baseline)
  Age, gender, education level, household income, employment status, marital status, language spoken, complete family history, current and previous illness and co-morbidities, and current medications
Oral Health Qualitative Interviews | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  using the German version of the "Oral Health Impact Profile" with 21 questions, score ranges from 0 to 21, high score Shows a low Quality of oral health, low score Shows a high Quality of life
Evaluation of inflammatory oral conditions | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  bleeding index (gingival bleeding index, bleeding on probing) in percentage, ranges from 0 to 100 %, optimal is less then 15 %
Evaluation of teeth related conditions | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  dental findings (attrition, bruxism, caries, dental implants, dentures, missing teeth, erosions, restorations (all classes))
Evaluation of Oral Fluids | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  crevicular fluid rate, salivary flow (stimulated, unstimulated)
Evaluation of periodontal attachment level | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  probing pocket depth, recessions, measuring in mm on 6 sites per tooth
Evaluation of oral hygiene | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  Plaque Index in %, ranges from 0 to 100%, less then 15 % Shows an optimal oral hygiene
Evaluation of periodontal status | Date of inclusion (baseline), after 8 weeks, after 16 weeks
  measuring with periodontal Screening index, ranges from 0 to 4, code 0 - oral health, 1-2 Gingivitis, 3-4 Periodontitis, additional findings as furcation involvement and loosening are documented

OTHER OUTCOMES:
Qualitative interviews in focus groups interviews | 16 weeks after inclusion
  Qualitative assessment will be carried out in 45-minute focus group interviews in 12 (randomized selected) patients participating in the study. The interviews will be recorded, transcribed and analyzed with qualitative content analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charite - Universitätsmedizin Berlin
Locations (1):
- Charite University, Berlin, Germany

REFERENCES:
- [Derived] Pappe CL, Lutzenberger S, Goebler K, Meier S, Jeitler M, Michalsen A, Dommisch H. Effect of a Whole-Food Plant-Based Diet on Periodontal Parameters in Patients With Cardiovascular Risk Factors: A Secondary Sub-Analysis of a Randomized Clinical Trial. J Clin Periodontol. 2025 Jan;52(1):125-136. doi: 10.1111/jcpe.14066. Epub 2024 Oct 14. PMID 39402877